CLINICAL TRIAL: NCT06716853
Title: An Open-label Phase 1/2 Study to Evaluate the Safety, Biological Response and Efficacy of a Single Dose of Temferon (Autologous CD34+-Enriched Hematopoietic Stem and Progenitors Cells Genetically Modified With Human Interferon-α2) in Patients With Metastatic Renal Cell Carcinoma
Brief Title: A Clinical Gene Therapy Study With Hematopoietic Stem Cells for the Treatment, With Single Dose of Temferon, of Patients Suffering From Metastatic Renal Cell Carcinoma
Acronym: TEM-GU
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Persistent challenges have been encountered in patient recruitment, difficulty in identifying a sufficient number of eligible subjects. The decision to terminate the study was not based on any safety concerns. Benefit-risk profile of IP unchanged.
Sponsor: Genenta Science (Industry)
Collaborators: Alira Health (Other); Arithmos srl (Unknown); Ospedale San Raffaele (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TEM-GU; 2024-512898-27-00 (EU CTIS Number)
Record Dates: First submitted 2024-11-15; First posted 2024-12-04 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Clear Cell RCC
Keywords: metastatic renal cell carcinoma; Temferon; Gene; Solid tumor; Immunotherapy
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — pembrolizumab; cabozantinib

STUDY DESIGN:
Intervention Model Description: This is an open label, single-centre phase 1/2 therapeutic-exploratory prospective study where Temferon will be administered to up to 12 patients split into two cohorts according to immune checkpoint inhibitor -ICI- therapy received in the six months prior to entry into the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab cohort (Experimental): At D+30 after Temferon, patients will start to receive pembrolizumab providing they have not received ICI in the 6 months prior to entry into the study. Patients allocated to pembrolizumab will receive pembrolizumab 400mg IV every 6 weeks commencing at D+30.
  Interventions: Genetic: Temferon; Biological: Pembrolizumab
- Cabozantinib cohort (Experimental): At D+30 after Temferon, in the event that a patient has received ICI in the 6 months prior to study entry and in case PD occurs (as assessed at D+30 or at subsequent visits), they will be receiving cabozantinib. Patients allocated to cabozantinib cohort will initiate treatment with 40mg QD
  Interventions: Genetic: Temferon; Drug: Cabozantinib

INTERVENTIONS:
Genetic: Temferon — Autologous CD34+-enriched hematopoietic progenitor cells exposed in vitro to specific lentiviral vector encoding for the human interferon-alpha 2 gene. Its expression is tightly controlled by the human TIE2 enhancer/promoter sequence and by a post-transcriptional regulation layer represented by target miRNA sequences. This enables suppression of interferon-alpha2 expression in HSPCs, thereby further increasing the specificity of the delivery strategy for their Tie2 expressing myeloid cell progeny.
Biological: Pembrolizumab — Pembrolizumab 400mg IV every 6 weeks commencing at D+30
  Arms: Pembrolizumab cohort
Drug: Cabozantinib — 40mg QD once PD occurs as assessed at D+30 or at subsequent visits
  Arms: Cabozantinib cohort

SUMMARY:
This is an open label, single-centre phase 1/2 study involving a single dose of Temferon, an investigational Advanced Therapy Medicinal Product (ATMP), to treat patients with metastatic clear cell renal cell carcinoma (RCC) with evidence of disease progression following at least two lines of standard of care (SoC) treatments.

DETAILED DESCRIPTION:
During Part A (Phase 1) of the study, Temferon will be administered to up to 12 patients, who are going to be split into two cohorts according to immune checkpoint inhibitor -ICI- therapy received in the six months prior to entry into the study, with a histologically confirmed diagnosis of metastatic RCC and evidence of disease progression following at least two lines of SoC treatments.

At D+30 after Temferon, patients will start to receive pembrolizumab providing they have not received ICI in the 6 months prior to entry into the study. Patients allocated to pembrolizumab will receive pembrolizumab 400mg IV every 6 weeks commencing at D+30.

In the event that a patient has received ICI in the 6 months prior to study entry, they will be allocated to the cabozantinib arm. Patients allocated to cabozantinib, will initiate treatment with 40mg QD once PD occurs as assessed at D+30 or at subsequent visits.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged between 18 - 70 years old
* Women of childbearing potential must have a negative pregnancy test at screening and agree to use two distinct acceptable methods of contraception (which may include partner contraception) for the duration of the study
* Men with partners of childbearing potential must be willing to use acceptable barrier contraceptive method during the trial or have undergone a vasectomy at least 6 months prior to study entry and confirmed by semen analysis
* Adequate cardiac, renal, hepatic, pulmonary, and hematologic function
* Patient able and willing to provide written informed consent and comply with study protocol and procedures
* Histologically confirmed diagnosis of unresectable, locally advanced/metastatic RCC with clear cell component, with or without sarcomatoid features
* Presence of a disease burden sufficiently large to permit biopsy
* Disease progression following approved standard of care treatments for metastatic disease
* ECOG PS 0-1
* Measurable disease at physical examination or at imaging assessment according to RECIST 1.1 criteria

Exclusion Criteria:

* Use of investigational agents or procedures in the 4 weeks prior to study enrolment (6 weeks for long-acting agents) or receipt of an experimental gene therapy product in the past 2 years
* History of current evidence of neuropsychiatric illness
* History of severe cardiovascular disease
* Evidence of haematological neoplasm
* Active alcohol or substance abuse within 6 months of the study
* Current pregnancy or lactation
* Expected to undergo a surgical intervention during the first 3 months of the study
* Known bleeding diathesis or history of abnormal/severe bleeding or any other known coagulation abnormalities that would contraindication a tissue biopsy, active treatment with anticoagulants.
* New CNS or rapidly growing metastases or carcinomatous meningitis
* Presence of hepatic metastases
* Previous allogenic bone marrow, renal, liver transplant
* Prior use of immunosuppressives in the previous 4 weeks prior to enrolment
* Clinically relevant active viral, bacterial or fungal infection
* Active autoimmune disease requiring disease modifying treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-10-22 (Actual); Primary Completion 2026-01-23 (Actual); Study Completion 2026-01-23 (Actual)

PRIMARY OUTCOMES:
Tolerability and safety of conditioning and Temferon, over the first 90 days following administration, as determined by the incidence of adverse events | First 90 days
  To assess tolerability and safety of conditioning and Temferon over the first 90 days following Temferon administration, as evaluated by the incidence of >=CTCAE Grade 2 adverse events.
Biological activity of Temferon, over the first 90 days following administration, as determined by the presence of Temferon-derived progeny in the tumor (IFN gene signature) | First 90 days
  To assess the biological activity of Temferon in the tumor of patients with metastatic renal cell carcinoma, over the first 90 days following Temferon administration, as determined by the change in IFN (interferon) gene signature in the tumor

SECONDARY OUTCOMES:
Long term tolerability and safety of Temferon as determined by the incidence of adverse events up to 1 year following Temferon administration according to CTCAE v5.0 criteria | 1 year following Temferon administration
Incidence, severity and duration of adverse events of special interest as indicated on the study protocol | Through study completion, an average of 1 year
Proportion of patients achieving hematological recovery by Day +30 | Day 30
Overall response rate per RECIST version 1.1 | RECIST criteria used at Screening, Baseline, Day +72, Day +120, Day +180, Day +210, Day +270, Day +360 or at any time disease progression or a secondary malignancy is suspected
  Defined as the proportion of patients who achieved a complete or partial response as their best overall response
Disease control rate following Temferon infusion | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale San Raffaele, Milan, Italy, Italy